CLINICAL TRIAL: NCT01714778
Title: Electronic Cigarettes: Potential Toxicant (Acrolein) and Nicotine Delivery in Users
Brief Title: Toxins and Delivery in e-Cigarette Users
Acronym: TADEUS
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: QMUL201208a
Record Dates: First submitted 2012-10-23; First posted 2012-10-26 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine is collected for analysis of a metabolite of acrolein (3-HPMA_.
  Blood is collected for analysis of nicotine.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- e-Cigarette: Smokers attempting to quit with behavioural support and e-Cigarettes.
  Interventions: Other: e-Cigarette

INTERVENTIONS:
Other: e-Cigarette

SUMMARY:
Electronic cigarettes or "e-cigarettes" (EC) may have a potential public health benefit as a safer alternative to smoking and possibly also as an aid in tobacco dependence treatment. However, there are concerns about their safety and whether they can deliver nicotine consistently and in doses necessary for such effects.

To be able to consider the safety of ECs and their potential in harm reduction, data are needed comparing the exposure to the potential toxicant, acrolein, in smokers of conventional cigarettes, users of EC, and people who use both products at the same time.

To accurately assess EC nicotine delivery, data are needed from people who use them regularly, as there is some evidence of higher and faster nicotine absorption in experienced users compared with naïve users who try them once in an artificial laboratory setting.

This study will provide information on both of these issues. Forty smokers will be given EC to use, in addition to behavioural support, as part of a stop smoking attempt. Levels of acrolein and nicotine will be measured before and after 4 weeks of EC use.

ELIGIBILITY:
Inclusion Criteria:

* Smokers who want help in quitting
* Aged 18 or over

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* People with any current serious illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Smokers from the community who wish to stop smoking.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in urinary 3HPMA levels after 4 weeks use of electronic cigarettes. | 4 weeks
  Change in urinary 3HPMA levels (a metabolite of acrolein) after 4 weeks use of electronic cigarettes, in both individuals who have stopped smoking conventional cigarettes and those who are still using them.

SECONDARY OUTCOMES:
Change in nicotine levels after 4 weeks use of electronic cigarettes (EC) | 4 weeks
  Change in blood nicotine levels obtained from using an EC after 4 weeks use of electronic cigarettes (10 participants only).
Electronic cigarette acceptability | 6 months
  Participants' views on electronic cigarettes
Use of electronic cigarettes | 6 months
  Participants' use of electronic cigarettes

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary University of London, London, United Kingdom